CLINICAL TRIAL: NCT01695070
Title: A Pilot Study of Maternally Administered Melatonin to Decrease the Level of Oxidative Stress in Human Pregnancies Affected by Intrauterine Growth Restriction.
Brief Title: Melatonin to Prevent Brain Injury in Unborn Growth Restricted Babies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Nicole Alers, MD, Monash University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1133-4541; ACTRN12612000858897 (Registry Identifier: Australian New Zealand Clinical Trial Registry)
Record Dates: First submitted 2012-09-07; First posted 2012-09-27 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melatonin (Experimental): Women with IUGR will take 4mg prolonged release melatonin oral tablets twice daily. Treatment will occur as soon as the diagnosis of intrauterine growth restriction is made and the patient has been enrolled to this study until birth. The overall duration of treatment will vary due to the nature of intrauterine growth restriction.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — 4mg prolonged release melatonin oral tablets twice daily
  Other Names: Circadin

SUMMARY:
Intrauterine growth restriction is the term used to describe a condition where an unborn baby does not reach its optimum size. In the short and long term, intrauterine growth restricted babies have a higher risk of serious disease and even death. It is well established that very low levels of oxygen in the baby's blood can harm the baby's health through a state known as oxidative stress. Currently, there is no established treatment available to treat intrauterine growth restriction or its complications. In experimental animal studies however, the naturally occuring hormone, melatonin, has been shown to significantly reduce oxidative stress and improve health of the unborn babies that have suffered from intrauterine growth restriction. This study aims to find out if the use melatonin twice per day throughout pregnancies affected by intrauterine growth restriction will lower the level of oxidative stress experienced by the unborn baby. If this is the case melatonin may help protect the unborn baby from damage caused by oxidative stress, this will be studied in a separate future study.

ELIGIBILITY:
Inclusion Criteria:

* Estimated fetal weight <10th percentile in combination with abnormal fetoplacental Doppler studies.
* Singleton pregnancy.
* Live fetus.
* Gestational age: from 23+0 weeks until 34+0 weeks.
* Normal fetal anatomy on ultrasound.
* Confirmed gestational age.
* No indication for immediate delivery.
* Basic understanding of the English language.
* 18 years or older.
* Consent obtained.

Exclusion Criteria:

* Fetal demise.
* Multiple pregnancy.
* Known abnormal karyotype.
* Presence of any congenital abnormality.
* Unknown duration of pregnancy.
* IUGR attributable to non-placental factors.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Oxidative stress in the umbilical artery | Once, at birth.
  Umbilical artery oxidative stress by measuring levels of malondialdehyde (MDA) and 8-isoprostane. Levels of MDA will be assessed using a Thiobarbituric Acid Reactive Substances Assay Kit (Cayman Chemical Item Number 10009055). Levels of 8-isoprostane will be assessed using an 8-Isoprostane Enzyme Immuno Assay Kit (Cayman Chemical Item Number 516351).

SECONDARY OUTCOMES:
Oxidative stress in maternal venous serum | Once within one week before start treatment and once per week during the treatment period (estimated to be an average of 4 weeks).
  Maternal serum oxidative stress will be assessed by measuring levels of malondialdehyde (MDA) and 8-isoprostane. Levels of MDA will be assessed using a Thiobarbituric Acid Reactive Substances Assay Kit (Cayman Chemical Item Number 10009055). Levels of 8-isoprostane will be assessed using an 8-Isoprostane Enzyme Immuno Assay Kit (Cayman Chemical Item Number 516351).
Fetoplacental Doppler studies | Once within one week before start treatment and twice per week during the treatment period (estimated to be an average of 4 weeks).
  Fetoplacental Doppler studies (umbilical artery, uterine artery, middle cerebral artery, ductus venosus). Fetoplacental Doppler studies are performed in the clinical assessment of women diagnosed with intrauterine growth restriction by sonography.
Placental oxidative stress | Once, at birth.
  Placental oxidative stress is assessed by measuring levels of malondialdehyde (MDA) and 8-isoprostane. Levels of MDA will be assessed using a Thiobarbituric Acid Reactive Substances Assay Kit (Cayman Chemical Item Number 10009055). Levels of 8-isoprostane will be assessed using an 8-Isoprostane Enzyme Immuno Assay Kit (Cayman Chemical Item Number 516351)
Gestational age at birth. | Once, at birth.
  Gestational age at birth will be calculated using the last menstrual period and ultrasound characteristics.
Composite neonatal outcome. | Participants will be followed for the duration of hospital stay, up to 12 months.
  Composite neonatal outcome (admission to NICU, duration of admission, need and duration of respiratory support, intraventricular haemorrhage, necrotising enterocolitis, abnormal neurological assessment, mortality before discharge). This composite neonatal outcome will be measured by collecting medical record data after clinical assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole O Alers, MD, Principal Investigator — The Ritchie Centre, Monash Institute of Medical Research, Monash University; Euan M Wallace, MBChB MD FRCOG FRANZCOG, Principal Investigator — Southern Health, The Ritchie Centre, Monash Institute of Medical Research, Monash University; Graham Jenkin, BSc PhD, Principal Investigator — The Ritchie Centre, Monash Institute of Medical Research; Suzanne L Miller, BSc PhD, Principal Investigator — The Ritchie Centre, Monash Institute of Medical Research
Locations (1):
- Southern Health: Monash Medical Centre and Jessie McPherson Private Hospital, Clayton, Victoria, Australia

REFERENCES:
- [Derived] Miller SL, Yawno T, Alers NO, Castillo-Melendez M, Supramaniam VG, VanZyl N, Sabaretnam T, Loose JM, Drummond GR, Walker DW, Jenkin G, Wallace EM. Antenatal antioxidant treatment with melatonin to decrease newborn neurodevelopmental deficits and brain injury caused by fetal growth restriction. J Pineal Res. 2014 Apr;56(3):283-94. doi: 10.1111/jpi.12121. Epub 2014 Feb 22. PMID 24456220
- [Derived] Alers NO, Jenkin G, Miller SL, Wallace EM. Antenatal melatonin as an antioxidant in human pregnancies complicated by fetal growth restriction--a phase I pilot clinical trial: study protocol. BMJ Open. 2013 Dec 23;3(12):e004141. doi: 10.1136/bmjopen-2013-004141. PMID 24366583